CLINICAL TRIAL: NCT04564352
Title: Hypolipidemic, Antioxidant Activity of Adansonia Digitata Juice Consumption
Brief Title: Hypolipidemic Effect of Adansonia Digitata
Acronym: AD
Status: Completed | Type: Observational
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, Ahmed M Ahmed, Associate professor of Clinical chemistry - college of Applied Medical Sciences - Taibah University, Taibah University
Other Study IDs: CLS 201978; Taibah University (Other: Deanship of scintific research)
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2: Adansonia digitata (Baobab)
  Interventions: Dietary Supplement: Adansonia digitata

INTERVENTIONS:
Dietary Supplement: Adansonia digitata — Juice of AD fruit
  Other Names: Baobab

SUMMARY:
Adansonia digitata L. (AD) also known as Baobab is a huge tree that grows in many countries in sub-Saharan Africa. Many studies talking about AD biological activity including hypolipidemic, antioxidant and antimicrobials in animal's but not in human, This study will be undertaken to examine the effect of AD juice consumption against lipid profiles in traditional users and blood samples will be collected form participant's for investigated of lipid profiles pre and post AD juice drinking and the results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Tradition users (drink AD juice)

Exclusion Criteria:

* Diabetes, hypertension, or chronic illness

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The study is association case-control in design and involved Sudanese adult subjects (>18 years old - 60 years) living in Saudi Arabia. The cases were subjects who use AD fruit juice as tradition juice.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Decrease cholesterol level | 6 month's
  Hypolipidemias

CONTACTS AND LOCATIONS:
Locations (1):
- Taibah University, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
After participant's allow us to share their data